CLINICAL TRIAL: NCT02603432
Title: A PHASE 3, MULTICENTER, MULTINATIONAL, RANDOMIZED, OPEN-LABEL, PARALLEL-ARM STUDY OF AVELUMAB (MSB0010718C) PLUS BEST SUPPORTIVE CARE VERSUS BEST SUPPORTIVE CARE ALONE AS A MAINTENANCE TREATMENT IN PATIENTS WITH LOCALLY ADVANCED OR METASTATIC UROTHELIAL CANCER WHOSE DISEASE DID NOT PROGRESS AFTER COMPLETION OF FIRST-LINE PLATINUM-CONTAINING CHEMOTHERAPY
Brief Title: A Study Of Avelumab In Patients With Locally Advanced Or Metastatic Urothelial Cancer (JAVELIN Bladder 100)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991001; 2015-003262-86 (EudraCT Number); JAVELIN BLADDER 100 (Other: Alias Study Number)
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Urothelial Cancer
Keywords: Bladder cancer; Urologic neoplasms; urothelial carcinoma; PD-L1; programmed cell death protein; maintenance treatment
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms; Carcinoma, Transitional Cell | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Avelumab plus Best Supportive Care (BSC)
  Interventions: Biological: Avelumab; Other: Best Supportive Care
- Arm B (Other): Best Supportive Care (BSC) alone
  Following the planned interim analysis for this study, eligible patients in Arm B whose cancer has not worsened and are still in the "watch and wait" part of the study will be given the option to receive Avelumab plus BSC. Prior to this, Arm B patients received BSC alone. All patients who choose not to receive Avelumab will be discontinued.
  Interventions: Other: Best Supportive Care; Biological: Following the planned interim analysis for this study: Avelumab

INTERVENTIONS:
Biological: Avelumab — 1 hour intravenous infusion every 2 weeks (Q2W) in 4 week cycles
  Arms: Arm A
Other: Best Supportive Care — BSC will be administered as deemed appropriate by the treating physician, and could include treatment with antibiotics, nutritional support, correction of metabolic disorders, optimal symptom control and pain management (including palliative radiotherapy), etc. BSC does not include any active anti-tumor therapy, however local radiotherapy of isolated lesions with palliative intent is acceptable.
Biological: Following the planned interim analysis for this study: Avelumab — 1 hour intravenous infusion every 2 weeks (Q2W) in 4 week cycles
  Arms: Arm B

SUMMARY:
The main purpose of this study is to compare maintenance treatment with avelumab plus best supportive care (BSC) with BSC alone, to determine if avelumab has an effect on survival in patients with locally advanced or metastatic urothelial cancer that did not worsen during or following completion of first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable locally advanced or metastatic transitional cell carcinoma of the urothelium
* Stage IV disease at the start of first-line chemotherapy
* Measurable disease (per RECIST v1.1) prior to the start of first-line chemotherapy
* Prior first-line chemotherapy must have consisted of at least 4 cycles and no more than 6 cycles of gemcitabine + cisplatin and/or gemcitabine + carboplatin
* No evidence of progressive disease following completion of first-line chemotherapy (i.e., ongoing CR, PR, or SD per RECIST v1.1 guidelines )

Exclusion Criteria:

* Prior adjuvant or neoadjuvant systemic therapy within 12 months of randomization
* Prior immunotherapy with IL-2, IFN-α, or an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA 4 antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Persisting toxicity related to prior therapy (Grade >1 NCI CTCAE v4.0); however, alopecia, sensory neuropathy (Grade 2 or less), or other (Grade 2 or less) adverse events not constituting a safety risk based on the investigator's judgement are acceptable.
* Patients with known symptomatic central nervous system (CNS) metastases requiring steroids
* Diagnosis of any other malignancy within 5 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast or of the cervix, low grade prostate cancer on surveillance without any plans for treatment intervention, or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (371):
- United States (16):
  - Anschutz Cancer Center Pavilion Pharmacy, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Colorado Denver, CTO (CTRC), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Cleveland Clinic Taussing Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Inova Schar Cancer Institute Infusion Pharmacy, Fairfax, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Argentina (6):
  - Centro de Investigacion Pergamino S.A., Pergamino, Buenos Aires
  - Fundación CENIT para la Investigación en Neurociencias, CABA
  - GP Diagnostico SRL, La Rioja
  - Hospital Regional Dr. Enrique Vera Barros, La Rioja
  - Instituto del Diagnostico, La Rioja
  - Centro Oncologico Riojano Integral (Cori), La Rioja
- Australia (49):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Concord Hospital, Concord, New South Wales
  - Dubbo Base Hospital, Dubbo, New South Wales
  - Ramsay Pharmacy, Kogarah, New South Wales
  - St George Private Hospital, Kogarah, New South Wales
  - Epic Pharmacy, Lismore, New South Wales
  - North Coast Radiology St Vincents, Lismore, New South Wales
  - Northern Rivers Pathology Service, Lismore, New South Wales
  - St Vincent's Pathology Lismore, Lismore, New South Wales
  - Macquarie Medical Imaging, Macquarie University, New South Wales
  - Macquarie University Hospital Pharmacy, Macquarie University, New South Wales
  - Macquarie University, Macquarie University, New South Wales
  - The Murwillumbah Hospital, Murwillubah, New South Wales
  - The Tweed Hospital Pharmacy Department, Tweed Heads, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - River City Pharmacy, Auchenflower, Queensland
  - Oncology Pharmacy, Birtinya, Queensland
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - The Townsville Hospital, Douglas, Queensland
  - Slade Health, Geebung, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Icon Cancer Care, South Brisbane, Queensland
  - Integrated Clinical Oncology Network (ICON) Corporate Office, South Brisbane, Queensland
  - Icon Cancer Care Southport, Southport, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - SA Pharmacy, Level 3 Pharmacy, Bedford Park, South Australia
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Cancer Care SA Pty Ltd, Kurralta Park, South Australia
  - Icon Cancer Care SA trading as Icon Pharmacy Adelaide, Kurralta Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - BHS Diagnostic Services, Ballarat, Victoria
  - Lake Imaging, Ballarat, Victoria
  - Ballarat Oncology & Haematology Services, Ballarat, Victoria
  - Box Hill Hospital - Pharmacy Department, Bulding B, Loading Dock (access via Thames St), Box Hill, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Eastern Health Clinical School, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Monash Medical Centre, East Bentleigh, Victoria
  - Moorabbin Radiology, East Bentleigh, Victoria
  - Ballarat Day Procedure Centre, Wendouree, Victoria
  - Ballarat Oncology & Haematology Services, Wendouree, Victoria
  - Nova Pharmacy, Wendouree, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God Murdoch Hospital, Murdoch, Western Australia
  - Slade Health, Mount Waverley
  - Macquarie Heart, New South Wales
- Belgium (7):
  - AZ Klina - Apotheek, Brasschaat
  - AZ Klina, Brasschaat
  - Hôpital Erasme, Brussels
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHU de Liège, Liège
  - GZA Sint-Augustinus, Wilrijk
- Brazil (21):
  - Hospital da Bahia, Salvador, Estado de Bahia
  - CENOB Centro de Oncologia da Bahia S/S Ltda. / Oncovida, Salvador, Estado de Bahia
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro, Rio de Janeiro
  - Associacao Hospital de Caridade Ijui, Ijuí, Rio Grande do Sul
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Associação Educadora São Carlos - AESC / Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Associação Educadora São Carlos - AESC / Hospital Mãe de Deus - Ambulatório Quimioterapia, Porto Alegre, Rio Grande do Sul
  - Associação Educadora São Carlos - AESC / Hospital Mãe de Deus - Centro de Abastecimento Farmaceut, Porto Alegre, Rio Grande do Sul
  - Associação Educadora São Carlos - AESC / Hospital Mãe de Deus - Farmácia Oncológica, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus/Aesc, Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia / Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundação FPio XII Barretos, Barretos, São Paulo
  - Fundação Pio XII Barretos, Barretos, São Paulo
  - Centro Integrado de Pesquisa Clinica - CIP, São José do Rio Preto, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Fundacao Faculdade de Medicina / Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sírio Libanês, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP - HCFMUSP, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein - SP, São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sírio Libanês/ Instituo Sirio Libanes de Ensino e Pesqu, São Paulo
- Canada (3):
  - William Osler Health System, Brampton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- Czechia (6):
  - Fakultni nemocnice u sv. Anny v Brne, Brno, Ceska Republika
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice u sv.Anny v Brne, Brno
  - Nemocnice Horovice, NH Hospital a.s., Hořovice
  - Nemocnice Horovice, Hořovice
- Denmark (13):
  - Aalborg Universitetshospital Syd, Aalborg
  - Aalborg Universitetshospital, Aalborg
  - Sygehusapoteket Aalborg, Aalborg
  - Aarhus Universitetshospital, Aarhus C
  - Aarhus Universitetshospital, Aarhus N
  - CT-Klinikken A/S, Aarhus N
  - Rigshospitalet, Onkologisk Klinik, afsnit 5073, Copenhagen OE
  - Herlev Hospital, Herlev
  - Herlev og Gentofte Hospital, Herlev
  - Klinik for Klinisk Fysiologi,Nuklearmedicin og PET, København Ø
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Odense
  - Odense Universitetshospital, Odense C
- France (30):
  - Groupe hospitalier Pitie Saleptriere, Paris, Cedex 13
  - Institut de cancérologie de l'Ouest - Site Paul Papin, Angers
  - Centre d'Oncologie et de Radiothérapie du Pays-Basque, Bayonne
  - Clinique CAPIO Belharra, Bayonne
  - CHU Besançon - Pharmacie Unite Essais cliniques, Besançon
  - CHU Besançon, Besançon
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Henri Mondor, Créteil
  - Hôpital Privé Toulon-Hyères - Clinique Sainte Marguerite, Hyères
  - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Centre Léon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital La Conception, Marseille
  - Hopital de La Timone, Marseille
  - CHU Nimes - Hopital Caremeau, Nîmes
  - CHU Nimes - Institut de Cancerologie du Gard, Nîmes
  - CHU Nimes, Nîmes
  - Groupe Hospitalier Pitié Salpêtrière, Paris
  - Centre Eugene Marquis, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHU de Rouen, Rouen
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest - Centre René Gauducheau, Saint-Herblain
  - Centre de Radiothérapie - Clinique Sainte Anne, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - Hopital Foch -Pharmacie, Suresnes
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Greece (6):
  - Medical Center of Athens, Marousi, Athens
  - Metropolitan General Hospital, Athens, PC
  - Sotiria General Chest Disease Hospital, Athens
  - Alexandra General Hospital, Oncology Department, Athens
  - University General Hospital of Patras, Division of Oncology, Pátrai
  - EUROMEDICA General Clinic of Thessaloniki, Thessaloniki
- Department of Clinical Oncology, Hong Kong, Hong Kong
- Hungary (2):
  - Kaposvári Egyetem Egészségügyi Centrum, Kaposvár
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
- India (6):
  - CIMS Cancer, Care Institute of Medical Sciences, CIMS Hospital, Ahmedabad, Gujarat
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Dr Ram Manohar Lohia (RML) Hospital & PGI MER, New Delhi, National Capital Territory of Delhi
  - Apollo Hospitals, Hyderabad, Telangana
  - Medica Superspecialty hospital, Kolkata, West Bengal
  - Rajiv Gandhi Cancer Institute And Research Centre, Delhi
- Israel (5):
  - Hadassah University Hospital, Kiryat Hadassah, Jerusalem
  - The Chaim Sheba Medical Center, Tel Litwinsky, Ramat - GAN
  - Assaf Harofe MC, Beer Yaakov
  - Rambam Health Care Campus, Haifa
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (35):
  - Farmacia Ospedaliera, Candiolo, (torino)
  - AOU Ospedali Riuniti di Ancona, Torrette, Ancona
  - U.O. Anatomia Patologica, Forlì, Forli-cesena
  - U.O. Radiologia, Forlì, Forli-cesena
  - U.O.S. Medicina Nucleare, Forlì, Forli-cesena
  - Farmacia Oncologica, Meldola, Forli-cesena
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Forli-cesena
  - U.O.C. Farmacia, Genova, Genoa
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Farmacia Studi Clinici, Rozzano, Milan
  - Istituto Clinico Humanitas, Rozzano, Milan
  - AUSL della Romagna - RAVENNA, Presidio Ospedaliero di Faenza, Faenza, Ravenna
  - Presidio Ospedaliero di Lugo, Lugo, Ravenna
  - Fondazione del Piemonte per l'Oncologia - IRCCS Candiolo, Candiolo, Torino
  - Farmacia Ospedaliera, Arezzo
  - Presidio Ospedaliero San Donato, Arezzo
  - Centro di Riferimento Oncologico - IRCCS, Aviano (PN)
  - S.O.C. di Farmacia, Aviano (PN)
  - Azienda Ospedaliero-Universitaria Policlinico S.Orsola Malpighi, Bologna
  - U.O. Farmacia Clinica - IDS, Bologna
  - Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan
  - SC Farmacia, Milan
  - Instituto Europeo di Oncologia, Milan
  - Servizio di Farmacia, Milan
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Naples
  - UOSC Farmacia, Naples
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, IRCCS Fondazione Giovanni Pascale, Napoli
  - S.C. Farmacia Ospedaliera, Napoli
  - A.O.U. Pisana Ospedale S. Chiara, Pisa
  - Presidio Ospedaliero di Ravenna, Ravenna
  - Servizio Farmacia Ospedaliera - Farmacia Oncologica, Ravenna
  - Azienda Ospedaliera San Camillo Forlanini_Oncologia Medica, Rome
  - U.O.C. Farmacia, Rome
  - Azienda Ospedaliera S. Maria di Terni, Terni
  - S.C. Farmacia Interna, Terni
- Japan (29):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University School of Medicine & Hospital, Hirosaki, Aomori
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - National Hospital Organization hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tsukuba Medical Center Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Kagoshima University Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka City University Hospital, Osaka
  - Tokushima University Hospital, Tokushima
  - Yamagata University Hospital, Yamagata
- Mexico (4):
  - Hospital Médica Campestre (Administradora Hospitalaria S.A de C.V.), León, Guanajuato
  - Centro de Investigación Clínica de Leon S.C., León, Guanajuato
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli, State of Mexico
- Netherlands (7):
  - Rijnstate Arnhem, Arnhem
  - Ziekenhuis Rijnstate, Arnhem
  - St Apotheek der Haarlemse Ziekenhuizen, Haarlem
  - Spaarne Gasthuis, Hoofddorp
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Radboudumc, Nijmegen
- New Zealand (5):
  - Auckland City Hospital Pharmacy, Grafton, Auckland
  - Auckland City Hospital, Grafton, Auckland
  - Slade Health Inward Goods, Auckalnd
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- Norway (6):
  - Akershus University Hospital, Lorenskog
  - Sykehusapoteket HF 23 Lørenskog, Lorenskog
  - Sykehusapoteket HF 23 Lørenskog, Nordbyhagen
  - Sykehusapoteket Lorenskog, Nordbyhagen
  - Bildediagnostisk avdeling, Nordbyhagen
  - Stavanger University Hospital, Stavanger
- Poland (7):
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw, Masovian Voivodeship
  - Centralny Szpital Kliniczny MSWiA, Warsaw, Masovian Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej im. Sw. Jana z Dukli, Lublin
  - Lecznice CITOMED Sp. z o.o., Torun
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu Szpital Obserwacyjno-Zakazny, Torun
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
  - Wojewodzki Szpital Zespolony im. L. Rydygiera, Szpital Specjalistyczny dla Dzieci I Doroslych, Torun
- Portugal (9):
  - Instituto Português de Oncologia de Coimbra Francisco Gentil, EPE, Coimbra
  - Hospital Da Luz Coimbra, SA, Coimbra
  - Centro Hospitalar de Lisboa Central, E.P.E. - Hospital de Santo António dos Capuchos, Lisbon
  - Hospital CUF Descobertas, SA, Lisbon
  - Dr. Campos Costa - Consultório de Tomografia Computorizada, S.A., Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de São João, EPE, Porto
  - Dr. Campos Costa - Consultório de Tomografia Computorizada, S.A.- Matosinhos, Senhora da Hora
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, EPE, Vila Real
- Russia (16):
  - State Budgetary Healthcare Insti. Republican Clinical Oncology Dispensary of the MoH of Bashk. Rep., Ufa, Bashkortostan Republic
  - Federal State Budgetary Institution "National medical research radiology center" MoH RF, Obninsk, Kaluga Oblast
  - Private Medical Institution "Evromedservice", Pushkin, Sankt-Peterburg
  - Principal Military Clinical Hospital n.a. N.N. Burdenko, Moscow
  - Moscow Research Oncology Institute named after P. A. Gertsen, Moscow
  - BHI of Omsk region "Clinical oncological dispensary", Omsk
  - FGBIH "Clinical Hospital #122 n.a. L.G. Sokolov of Federal Medico-biological agency", Saint Petersburg
  - Non-State Healthcare Institution "Railway Clinical Hospital JSC RZhD", Saint Petersburg
  - FSBEI HE "First St. Petersburg State Medical University n. a. academician l.P Pavlov" MoH RF, Saint Petersburg
  - FSBEI HE "First St. Petersburg State Medical University n.a. academician I.P Pavlov" MoH RF, Saint Petersburg
  - FSBEI HE "First St. Petersburg State Medical University n.a. academician I.P Pavlov", Saint Petersburg
  - "Ramsay Diagnostics Rus", LLC, Saint Petersburg
  - FSBI "Russian Scientific Center For Radiology and Surgical Technologies n.a. Academician A.M. Granov, Saint Petersburg
  - Hospital Orkli, LLC, Saint Petersburg
  - Mart, Llc, Saint Petersburg
  - SHI YR "Regional Clinical Oncology Hospital", Yaroslavl
- Serbia (3):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Clinical Centre Nis, Clinic of Oncology, Niš
- South Korea (11):
  - National Cancer Center - Clinical Trial Pharmacy, Goyang-si, Gyeonggi-do
  - National Cancer Center Urology center for Prostate Cancer, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Clinical Pharmacy, Seongnam-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Chungnam National University Hospital, Clinical Pharmacy, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center - Clinical Trial Pharmacy, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center Clinical Trial Pharmacy, Seoul
  - Samsung Medical Center, Seoul
- Spain (50):
  - C.H. Univ. Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Comarcal General de Elda de Virgen de la Salud, Elda, Alicante
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catalá d'Oncología - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Institut Catalá d'Oncología, L'Hospitalet de Llobregat, Barcelona
  - Althaia. Xarxa Assistencial Universitaria de Manresa, Manresa, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - C. H. Universitario de Vigo- Hospital Álvaro Cunqueiro, Vigo, Galicia
  - C.H. Universitario de Vigo- Hospital Meixoeiro, Vigo, Galicia
  - Hospital Universitario Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Elche, Elche, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Vithas Internacional Medimar, Alicante
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Quiron of Barcelona, Barcelona
  - Hospital Quiron, Barcelona
  - Hospital Quirón de Barcelona, Barcelona
  - Hospital de La Santa Creu i Sant pau_Oncology department, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - CETIR Grup Medic, Barcelona
  - Cetir, Centre Mèdic, S.L, Barcelona
  - Hospital de Vall d'Hebron, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Laboratorio Dr. F. Echevarne Analisis, S.A, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Reina Sofía, Córdoba
  - H. univ Girona Dr. Josep Trueta - lnstitut Catala d'Oncologia, Girona
  - Institut Catala d'Oncologia, Girona
  - Institut Diagnostic de la lmatge, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Fundacion Maria Rafols para la investigacion del Diagnostico de la imagen, Madrid
  - Gabinete Radiologico Doctor Pita, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Ruber International, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - APL, Stockholm
  - Karolinska University Hospital, Stockholm
- Taiwan (10):
  - Clinical Trial Pharmacy, China Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Department of Pharmacy, National Cheng Kung University Hospital, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Investigational Drug services, National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Pharmacy, Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
  - Chemotherapy pharmacy, Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (6):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - St Bartholomew 's Hospital, Barts Health NHS Trust, London
  - St. Bartholomew's Hospital, Barts Health NHS Trust, London
  - Guy's & St. Thomas' NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, Guy's Hospital, London
  - Churchill Hospital, Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Vashistha R, Noor Z, Dasgupta S, Pu J, Deng S. Application of statistical machine learning in biomarker selection. Sci Rep. 2023 Oct 26;13(1):18331. doi: 10.1038/s41598-023-45323-9. PMID 37884606
- [Derived] Bellmunt J, Chang J, Pavilack-Kirker M, Cappelleri JC, Costa N, Esterberg E, Kearney M, Hitchens A, Candrilli SD, Ajmera M. Evaluating Real-World Characteristics of Patients With Advanced Urothelial Carcinoma Eligible for Avelumab Maintenance Therapy: A Multicountry Retrospective Medical Chart Review. Clin Genitourin Cancer. 2023 Aug;21(4):459-466. doi: 10.1016/j.clgc.2023.03.011. Epub 2023 Mar 31. PMID 37149458
- [Derived] Grivas P, Park SH, Voog E, Caserta C, Gurney H, Bellmunt J, Kalofonos H, Ullen A, Loriot Y, Sridhar SS, Yamamoto Y, Petrylak DP, Sternberg CN, Gupta S, Huang B, Costa N, Laliberte RJ, di Pietro A, Valderrama BP, Powles T. Avelumab First-line Maintenance Therapy for Advanced Urothelial Carcinoma: Comprehensive Clinical Subgroup Analyses from the JAVELIN Bladder 100 Phase 3 Trial. Eur Urol. 2023 Jul;84(1):95-108. doi: 10.1016/j.eururo.2023.03.030. Epub 2023 Apr 28. PMID 37121850
- [Derived] Powles T, Park SH, Caserta C, Valderrama BP, Gurney H, Ullen A, Loriot Y, Sridhar SS, Sternberg CN, Bellmunt J, Aragon-Ching JB, Wang J, Huang B, Laliberte RJ, di Pietro A, Grivas P. Avelumab First-Line Maintenance for Advanced Urothelial Carcinoma: Results From the JAVELIN Bladder 100 Trial After >/=2 Years of Follow-Up. J Clin Oncol. 2023 Jul 1;41(19):3486-3492. doi: 10.1200/JCO.22.01792. Epub 2023 Apr 18. PMID 37071838
- [Derived] Lee JL, Desai C, Park SH, Tsuchiya N, Su PJ, Chan TTW, Gurney H, Gao S, Wang J, Sandner R, di Pietro A, Eto M. Avelumab first-line maintenance plus best supportive care (BSC) vs. BSC alone for advanced urothelial carcinoma: JAVELIN Bladder 100 Asian subgroup analysis. Urol Oncol. 2023 May;41(5):256.e17-256.e25. doi: 10.1016/j.urolonc.2023.02.002. Epub 2023 Apr 3. PMID 37019764
- [Derived] Grivas P, Kopyltsov E, Su PJ, Parnis FX, Park SH, Yamamoto Y, Fong PC, Tournigand C, Climent Duran MA, Bamias A, Caserta C, Chang J, Cislo P, di Pietro A, Wang J, Powles T. Patient-reported Outcomes from JAVELIN Bladder 100: Avelumab First-line Maintenance Plus Best Supportive Care Versus Best Supportive Care Alone for Advanced Urothelial Carcinoma. Eur Urol. 2023 Apr;83(4):320-328. doi: 10.1016/j.eururo.2022.04.016. Epub 2022 May 30. PMID 35654659
- [Derived] Powles T, Park SH, Voog E, Caserta C, Valderrama BP, Gurney H, Kalofonos H, Radulovic S, Demey W, Ullen A, Loriot Y, Sridhar SS, Tsuchiya N, Kopyltsov E, Sternberg CN, Bellmunt J, Aragon-Ching JB, Petrylak DP, Laliberte RJ, Huang B, Costa N, Blake-Haskins JA, Grivas P. Plain language summary of results from the JAVELIN Bladder 100 study: avelumab maintenance treatment for advanced urothelial cancer. Future Oncol. 2022 Jun;18(19):2361-2371. doi: 10.2217/fon-2021-1631. Epub 2022 Apr 13. PMID 35416053
- [Derived] Tomita Y, Yamamoto Y, Tsuchiya N, Kanayama H, Eto M, Miyake H, Powles T, Yoshida M, Koide Y, Umeyama Y, di Pietro A, Uemura H. Avelumab first-line maintenance plus best supportive care (BSC) vs BSC alone for advanced urothelial carcinoma: JAVELIN Bladder 100 Japanese subgroup analysis. Int J Clin Oncol. 2022 Feb;27(2):383-395. doi: 10.1007/s10147-021-02067-8. Epub 2022 Jan 1. PMID 34973108
- [Derived] Powles T, Sridhar SS, Loriot Y, Bellmunt J, Mu XJ, Ching KA, Pu J, Sternberg CN, Petrylak DP, Tambaro R, Dourthe LM, Alvarez-Fernandez C, Aarts M, di Pietro A, Grivas P, Davis CB. Avelumab maintenance in advanced urothelial carcinoma: biomarker analysis of the phase 3 JAVELIN Bladder 100 trial. Nat Med. 2021 Dec;27(12):2200-2211. doi: 10.1038/s41591-021-01579-0. Epub 2021 Dec 10. PMID 34893775
- [Derived] Powles T, Park SH, Voog E, Caserta C, Valderrama BP, Gurney H, Kalofonos H, Radulovic S, Demey W, Ullen A, Loriot Y, Sridhar SS, Tsuchiya N, Kopyltsov E, Sternberg CN, Bellmunt J, Aragon-Ching JB, Petrylak DP, Laliberte R, Wang J, Huang B, Davis C, Fowst C, Costa N, Blake-Haskins JA, di Pietro A, Grivas P. Avelumab Maintenance Therapy for Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2020 Sep 24;383(13):1218-1230. doi: 10.1056/NEJMoa2002788. Epub 2020 Sep 18. PMID 32945632
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included only those participants who did not show evidence of disease progression after completion of at least 4 and not more than 6 cycles of first-line platinum-containing chemotherapy (prior to this study).
Groups:
- Avelumab + Best Supportive Care (BSC): Participants received an intravenous (IV) infusion of 10 milligrams per kilograms (mg/kg) of Avelumab along with BSC, on Day 1 and 15 of each 28 days treatment cycle, until confirmed disease progression, participant refusal, lost to follow up, unacceptable toxicity, or study termination by the sponsor, whichever occurred first. BSC was administered as per the treating physician. Participants were followed up until death, end of the study or withdrawal of consent, whichever comes first, regardless of initiation of new anti-cancer therapy.
- Best Supportive Care: As prescribed by the treating physician, participants received BSC which included treatment with antibiotics, nutritional support, correction of metabolic disorders, optimal symptom control and pain management, until confirmed disease progression, participant refusal, lost to follow up, unacceptable toxicity, or study termination by the sponsor, whichever occurred first. Participants were followed up until death, end of the study or withdrawal of consent, whichever comes first, regardless of initiation of new anti-cancer therapy.
Period: Overall Study
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Started | 350 | 350
Completed | 16 | 1
Not Completed | 334 | 349
Not completed — Adverse Event | 1 | 0
Not completed — Death | 221 | 242
Not completed — Lost to Follow-up | 3 | 9
Not completed — Progressive Disease | 7 | 5
Not completed — Withdrawal by Subject | 12 | 18
Not completed — No Longer Meets Eligibility Criteria | 3 | 0
Not completed — Study terminated by sponsor | 74 | 75
Not completed — Other | 13 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care | Total
Number analyzed (Participants) | 350 | 350 | 700
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.20 (9.52) | 67.7 (9.20) | 67.44 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 75 | 159
  Male | 266 | 275 | 541
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 12 | 30
  Not Hispanic or Latino | 286 | 298 | 584
  Unknown or Not Reported | 46 | 40 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 75 | 81 | 156
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 232 | 238 | 470
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 41 | 31 | 72

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time (in months) from the date of randomization to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From randomization to discontinuation from the study, death or date of censoring, whichever occurred first (for a maximum duration of 41 months)
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
months | 21.4 [18.9 to 26.1] | 14.3 [12.9 to 17.9]
Statistical Analysis 1: Comparison: Avelumab + Best Supportive Care (BSC) vs Best Supportive Care; Test type: Superiority; p = 0.0005, Log Rank — One-sided log-rank test was used; Analysis was performed using a Cox's Proportional Hazard model; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.556 to 0.863]

2. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR)
Description: BICR assessed PFS: Duration from randomization until disease progression (PD) or death. PD as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 was defined for target disease as at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (included baseline sum if that was smallest on study). In addition to relative increase of 20%, sum must have also demonstrated an absolute increase of at least 5 millimeters. For non-target disease: PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy. Appearance of any new unequivocal malignant lesion was also considered PD. Analysis was performed using Kaplan-Meier. PFS data was censored on date of last adequate tumor assessment for participants with no event (PD or death), who started new anti-cancer therapy prior to an event or with an event after 2 or more missing tumor assessments.
Time Frame: From randomization to date of progression of disease, discontinuation from the study, death or date of censoring, whichever occurred first (for a maximum duration of 41 months)
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
months | 3.7 [3.5 to 5.5] | 2.0 [1.9 to 2.7]

3. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by Investigator
Description: Investigator assessed PFS: Duration from randomization to first documentation of PD or death, whichever occurred first. PD as per RECIST version 1.1 was defined for target disease as at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (this included baseline sum if that was smallest on study). In addition to relative increase of 20%, sum must have also demonstrated an absolute increase of at least 5 mm. For non-target disease: PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy. Appearance of any new unequivocal malignant lesion was also considered PD. Analysis was performed using Kaplan-Meier. PFS data was censored on date of last adequate tumor assessment for participants with no event (PD or death), who started a new anti-cancer therapy prior to an event or with an event after 2 or more missing tumor assessments.
Time Frame: as for outcome 2
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
months | 5.5 [4.2 to 7.2] | 2.1 [1.9 to 3.0]

4. Secondary Outcome: Percentage of Participants With Objective Response (OR) as Assessed by Blinded Independent Central Review (BICR)
Description: BICR assessed objective response according to RECIST version 1.1, was defined as participants with confirmed best overall response of complete response (CR) or partial response (PR). CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions.
Time Frame: From randomization to progression of disease, start of new anti-cancer therapy or discontinuation from study or death, whichever occurred first (for a maximum duration of 41 months)
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
percentage of participants | 9.7 [6.8 to 13.3] | 1.4 [0.5 to 3.3]

5. Secondary Outcome: Percentage of Participants With Objective Response as Assessed by Investigator
Description: Investigator assessed objective response according to RECIST version 1.1, was defined as participants with confirmed best overall response of CR or PR. CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. A CR also required normalization of tumor marker levels and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions.
Time Frame: as for outcome 4
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
percentage of participants | 12.3 [9.0 to 16.2] | 3.4 [1.8 to 5.9]

6. Secondary Outcome: Time to Tumor Response (TTR) as Assessed by Blinded Independent Central Review (BICR)
Description: TTR was defined, for participants with an objective response as the time from 'start date' to the first documentation of objective tumor response (CR or PR), which was confirmed subsequently. CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions.
Time Frame: From the date of randomization to the first documentation of objective response (CR or PR) (for a maximum duration of 41 months)
Population: The full analysis set included all randomized participants. Here, 'Overall Number of participants analyzed (N)' signifies participants who were evaluable for this outcome measure (OM).
Measure: Median (Full Range); unit: months
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 34 | 5
months | 2.0 [1.7 to 16.4] | 2.0 [1.8 to 7.0]

7. Secondary Outcome: Time to Tumor Response (TTR) as Assessed by Investigator
Description: TTR was defined, for participants with an objective response as the time from 'start date' to the first documentation of objective tumor response (CR or PR). CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. A CR also required normalization of tumor marker levels and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions.
Time Frame: as for outcome 6
Population: The full analysis set included all randomized participants. Here, 'Overall Number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 43 | 12
months | 2.0 [1.8 to 22.2] | 1.9 [1.1 to 10.9]

8. Secondary Outcome: Duration of Response (DOR) as Assessed by Blinded Independent Central Review (BICR)
Description: BICR assessed DOR: time from first documentation of OR (confirmed CR or PR) to date of first documentation of PD or death due to any cause. As per RECIST version 1.1, CR: complete disappearance of all target and non-target lesions, with exception of nodal disease sustained for 4 weeks. Any pathological lymph nodes reduced in short axis to <10 mm. PR: at least 30% decrease in sum of longest dimensions of target lesions taking as reference baseline sum longest dimensions. PD for target disease: at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study and relative increase of 20%, sum also demonstrated absolute increase of at least 5 mm. PD for non-target disease: unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy. Appearance of any new unequivocal malignant lesion was also considered PD.
Time Frame: First response subsequently confirmed to progression of disease or start of new anti-cancer therapy or discontinuation from the study or death, whichever occurred first (for a maximum duration of 41 months)
Population: Analysis was performed on subset of randomized participants, who had objective response, as assessed by BICR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 34 | 5
months | NA [15.6 to NA] — Median and upper limit of 95% Confidence Interval (CI) were not estimable due to limited number of events. | NA [NA to NA] — Median and 95% CI were not estimable due to limited number of events.

9. Secondary Outcome: Duration of Response (DOR) as Assessed by Investigator
Description: Investigator assessed DOR: time from first documentation of OR (confirmed CR or PR) to date of first documentation of PD or death due to any cause. As per RECIST version 1.1, CR: complete disappearance of all target and non-target lesions, with exception of nodal disease sustained for 4 weeks. Additionally, normalization of tumor marker levels and any pathological lymph nodes reduced in short axis to <10 mm. PR: at least 30% decrease in sum of longest dimensions of target lesions taking as reference baseline sum longest dimensions. PD for target disease: at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study and relative increase of 20%, sum also demonstrated absolute increase of at least 5 mm. PD for non-target disease: unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy. Appearance of any new unequivocal malignant lesion was also considered PD.
Time Frame: as for outcome 8
Population: Analysis was performed on subset of randomized participants, who had objective response, as assessed by Investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 43 | 12
months | 25.6 [12.0 to NA] — The upper limit of 95% CI was not estimable due to limited number of events. | NA [3.6 to NA] — Median and upper limit of 95% CI were not estimable due to limited number of events.

10. Secondary Outcome: Percentage of Participants With Disease Control (DC) as Assessed by Blinded Independent Central Review (BICR)
Description: Disease Control (DC) was defined as a best overall response of CR, PR, non-CR/non-PD or stable disease (SD) as assessed by BICR. CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. Non-CR/Non-PD was defined as persistence of any non-target lesions and/or tumor marker level above the normal limits. SD was defined as not to qualify for CR, PR or PD for target lesions and followed PR only if the sum increased by less than 20% from the nadir, but enough that a previously documented 30% decrease no longer holds.
Time Frame: From randomization to PD, death or start of new anti-cancer therapy (for a maximum duration of 41 months)
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
percentage of participants | 41.1 [35.9 to 46.5] | 27.4 [22.8 to 32.4]

11. Secondary Outcome: Percentage of Participants With Disease Control (DC) as Assessed by Investigator
Description: DC was defined as a best overall response of CR, PR, non-CR/non-PD or SD as assessed by Investigator. CR was defined as complete disappearance of all target and non-target lesions, with the exception of nodal disease and sustained for at least 4 weeks. Additionally, normalization of tumor marker levels and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least 30% decrease in the sum of the longest dimensions of target lesions taking as reference the baseline sum longest dimensions. Non-CR/Non-PD was defined as persistence of any non-target lesions and/or tumor marker level above the normal limits. SD was defined as not to qualify for CR, PR or PD for target lesions and followed PR only if the sum increased by less than 20% from the nadir, but enough that a previously documented 30% decrease no longer holds.
Time Frame: From randomization to PD, death or start of new anti-cancer therapy (for a maximum duration of 41 months)
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
percentage of participants | 50.9 [45.5 to 56.2] | 34.0 [29.0 to 39.2]

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) Graded Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03, Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Treatment-emergent AEs are events between first dose of study drug and up to 90 days after last dose of study drug or end of treatment (EOT) visit, that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: For "Avelumab + Best Supportive Care (BSC)'' group: Day1 up to 90 days after last dose of study drug; for BSC group: Day1 up to 90 days after EOT visit (for a maximum duration of up to approximately 70 months for both groups)
Population: Safety analysis set included all participants who had received at least one dose of study drug on arm 'Avelumab+BSC' or completed Cycle 1 Day (C1D1) on arm 'BSC'.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 344 | 345
Participants
  Grade 1 | 37 | 76
  Grade 2 | 113 | 104
  Grade 3 | 163 | 58
  Grade 4 | 18 | 8
  Grade 5 | 7 | 24

13. Secondary Outcome: Number of Participants With Laboratory Abnormalities Greater Than or Equal to (>=) Grade 3 (G3), Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: Hematology (Anemia G3: hemoglobin<8.0 grams per deciliter [g/dL],<4.9 millimoles (mmol)/liter (L),<80 g/L, transfusion indicated, Grade 4 [G4]: life-threatening consequences, urgent intervention indicated, Grade 5 [G5]: death; platelet count decreased-G3:<50.0 to 25.0*10^9/L, G4: <25.0*10^9/L; lymphocyte count decreased-G3:<0.5-0.2*10^9/L, G4:<0.2*10^9/L; neutrophil count decreased-G3:<1.0 to 0.5*10^9 /L, G4:<0.5*10^9/L). Chemistry (creatinine increased-G3:>3.0 to 6.0*upper limit of normal [ULN], G4:>6.0*ULN; serum amylase increased, lipase increased-G3:>2.0- 5.0*ULN, G4:>5.0*ULN. Aspartate aminotransferase [AST], alanine aminotransferase [ALT]-G3:>5.0 to 20.0*ULN, G4:>20.0*ULN]. Blood bilirubin increased-[G3:>3.0 to 10.0*ULN, G4:>10.0*ULN], Creatine phosphokinase [CPK] increased- [G3:>5.0 to 10.0*ULN, G4:>10.0*ULN], Hyperglycemia-[G3:>250 to 500 mg/dL; >13.9 to 27.8 mmol/L hospitalization indicated, G4:>500 mg/DL; >27.8 mmol/L life-threatening consequences]).
Time Frame: as for outcome 12
Population: Safety analysis set included all participants who had received at least one dose of study drug on arm 'Avelumab+BSC' or completed C1D1 on arm 'BSC'. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number analyzed (n)' = Participants evaluable for this outcome measure for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 344 | 345
Participants
  Anemia: number analyzed (Participants) | 344 | 339
  Anemia | 16 | 12
  Platelet Count Decreased: number analyzed (Participants) | 344 | 339
  Platelet Count Decreased | 3 | 1
  Lymphocyte Count Decreased: number analyzed (Participants) | 344 | 339
  Lymphocyte Count Decreased | 20 | 11
  Neutrophil Count Decreased: number analyzed (Participants) | 344 | 339
  Neutrophil Count Decreased | 7 | 0
  Creatinine Increased: number analyzed (Participants) | 344 | 341
  Creatinine Increased | 7 | 5
  Serum Amylase Increased: number analyzed (Participants) | 340 | 329
  Serum Amylase Increased | 25 | 9
  Lipase Increased: number analyzed (Participants) | 343 | 332
  Lipase Increased | 37 | 22
  ALT Increased: number analyzed (Participants) | 344 | 341
  ALT Increased | 11 | 3
  AST Increased: number analyzed (Participants) | 344 | 340
  AST Increased | 6 | 3
  Blood Bilirubin Increased: number analyzed (Participants) | 344 | 340
  Blood Bilirubin Increased | 0 | 3
  CPK Increased: number analyzed (Participants) | 339 | 331
  CPK Increased | 9 | 0
  Hyperglycemia: number analyzed (Participants) | 344 | 341
  Hyperglycemia | 28 | 16

14. Secondary Outcome: Change From Baseline in Vital Signs - Blood Pressure at Day 1 of Cycle 2, 3, 4, 5, 6, 7 and End of Treatment (EOT) Visit
Description: Vital signs included blood pressure and pulse rate. Blood pressure included sitting diastolic blood pressure (DBP) and sitting systolic blood pressure (SBP).
Time Frame: Baseline (Day [D] 1 of Cycle [C] 1), Day 1 of Cycle 2, 3, 4, 5, 6, 7 , EOT visit (for a maximum duration of 41 months) (each cycle=28 days)
Population: Safety set analyzed. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 344 | 345
millimeters of mercury
  Baseline (C1D1): Sitting DBP: number analyzed (Participants) | 324 | 329
  Baseline (C1D1): Sitting DBP | 75.7 (10.81) | 77.0 (10.48)
  Change at Cycle 2, Day 1: Sitting DBP: number analyzed (Participants) | 295 | 287
  Change at Cycle 2, Day 1: Sitting DBP | -0.9 (9.37) | -0.0 (9.06)
  Change at Cycle 3, Day 1: Sitting DBP: number analyzed (Participants) | 268 | 228
  Change at Cycle 3, Day 1: Sitting DBP | -1.7 (10.36) | -1.6 (9.38)
  Change at Cycle 4, Day 1: Sitting DBP: number analyzed (Participants) | 230 | 153
  Change at Cycle 4, Day 1: Sitting DBP | -1.7 (9.97) | -1.0 (9.90)
  Change at Cycle 5, Day 1: Sitting DBP: number analyzed (Participants) | 201 | 119
  Change at Cycle 5, Day 1: Sitting DBP | -1.1 (10.60) | -1.0 (10.22)
  Change at Cycle 6, Day 1: Sitting DBP: number analyzed (Participants) | 181 | 107
  Change at Cycle 6, Day 1: Sitting DBP | -1.2 (10.89) | -1.1 (10.89)
  Change at Cycle 7, Day 1: Sitting DBP: number analyzed (Participants) | 158 | 81
  Change at Cycle 7, Day 1: Sitting DBP | -0.7 (10.90) | 0.2 (9.95)
  Change at End of Treatment: Sitting DBP: number analyzed (Participants) | 190 | 237
  Change at End of Treatment: Sitting DBP | -0.1 (12.09) | -1.7 (10.23)
  Baseline (C1D1): Sitting SBP: number analyzed (Participants) | 324 | 329
  Baseline (C1D1): Sitting SBP | 131.3 (17.34) | 130.6 (16.32)
  Change at Cycle 2, Day 1: Sitting SBP: number analyzed (Participants) | 295 | 287
  Change at Cycle 2, Day 1: Sitting SBP | -2.2 (14.85) | -0.3 (13.79)
  Change at Cycle 3, Day 1: Sitting SBP: number analyzed (Participants) | 268 | 228
  Change at Cycle 3, Day 1: Sitting SBP | -1.9 (16.10) | 1.0 (14.94)
  Change at Cycle 4, Day 1: Sitting SBP: number analyzed (Participants) | 230 | 153
  Change at Cycle 4, Day 1: Sitting SBP | -0.6 (16.54) | 1.3 (16.54)
  Change at Cycle 5, Day 1: Sitting SBP: number analyzed (Participants) | 201 | 119
  Change at Cycle 5, Day 1: Sitting SBP | -1.9 (15.49) | 1.9 (15.85)
  Change at Cycle 6, Day 1: Sitting SBP: number analyzed (Participants) | 181 | 107
  Change at Cycle 6, Day 1: Sitting SBP | -2.3 (15.77) | 3.3 (16.81)
  Change at Cycle 7, Day 1: Sitting SBP: number analyzed (Participants) | 158 | 81
  Change at Cycle 7, Day 1: Sitting SBP | -1.8 (16.13) | 2.7 (19.86)
  Change at End of Treatment: Sitting SBP: number analyzed (Participants) | 190 | 237
  Change at End of Treatment: Sitting SBP | -0.9 (18.99) | -0.3 (16.78)

15. Secondary Outcome: Change From Baseline in Vital Signs - Pulse Rate at Day 1 of Cycle 2, 3, 4, 5, 6, 7 and End of Treatment (EOT) Visit
Description: Vital signs included blood pressure and pulse rate. Changes from baseline in sitting pulse rate were summarized.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 344 | 345
beats per minute
  Baseline (C1D1): number analyzed (Participants) | 324 | 327
  Baseline (C1D1) | 76.1 (12.84) | 77.1 (12.95)
  Change at Cycle 2, Day 1: number analyzed (Participants) | 295 | 286
  Change at Cycle 2, Day 1 | 0.3 (11.81) | 0.1 (9.98)
  Change at Cycle 3, Day 1: number analyzed (Participants) | 268 | 226
  Change at Cycle 3, Day 1 | -0.2 (12.10) | -0.4 (10.20)
  Change at Cycle 4, Day 1: number analyzed (Participants) | 230 | 152
  Change at Cycle 4, Day 1 | -0.5 (12.84) | -0.1 (11.26)
  Change at Cycle 5, Day 1: number analyzed (Participants) | 201 | 118
  Change at Cycle 5, Day 1 | 0.4 (12.32) | -1.0 (11.45)
  Change at Cycle 6, Day 1: number analyzed (Participants) | 181 | 105
  Change at Cycle 6, Day 1 | -0.8 (11.54) | -2.6 (10.52)
  Change at Cycle 7, Day 1: number analyzed (Participants) | 158 | 80
  Change at Cycle 7, Day 1 | -0.6 (11.89) | -2.6 (11.48)
  Change at End of Treatment: number analyzed (Participants) | 190 | 235
  Change at End of Treatment | 2.5 (12.25) | 1.4 (12.45)

16. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Avelumab
Description: The Lower Limit of Quantitation (LLQ) of avelumab was 0.20 micrograms (mcg)/milliliter (mL). Data for this outcome measure was not collected for reporting group "Best Supportive Care", since avelumab was not administered in this arm.
Time Frame: End of avelumab infusion on Day 1 of Cycle 1, 2, 3, 5, 7, 9, 11, 13 and Day 15 of Cycle 1, 2, 3 (each cycle=28 days)
Population: Avelumab pharmacokinetic (PK) parameter analysis set: all participants who received at least one dose of avelumab and who had at least one post-dose concentration measurement above the LLQ for avelumab. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'n' signifies participants evaluable for this OM at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Avelumab + Best Supportive Care (BSC)
Number analyzed (Participants) | 344
microgram per milliliter (mcg/mL)
  Cycle 1, Day 1: number analyzed (Participants) | 295
  Cycle 1, Day 1 | 192.7 (68.4)
  Cycle 1, Day 15: number analyzed (Participants) | 283
  Cycle 1, Day 15 | 216.2 (49.6)
  Cycle 2, Day 1: number analyzed (Participants) | 274
  Cycle 2, Day 1 | 201.5 (54.5)
  Cycle 2, Day 15: number analyzed (Participants) | 262
  Cycle 2, Day 15 | 208.5 (60.2)
  Cycle 3, Day 1: number analyzed (Participants) | 251
  Cycle 3, Day 1 | 213.1 (39.6)
  Cycle 3, Day 15: number analyzed (Participants) | 228
  Cycle 3, Day 15 | 213.1 (52.7)
  Cycle 5, Day 1: number analyzed (Participants) | 179
  Cycle 5, Day 1 | 197.5 (67.7)
  Cycle 7, Day 1: number analyzed (Participants) | 147
  Cycle 7, Day 1 | 191.9 (86.2)
  Cycle 9, Day 1: number analyzed (Participants) | 111
  Cycle 9, Day 1 | 168.9 (84.4)
  Cycle 11, Day 1: number analyzed (Participants) | 86
  Cycle 11, Day 1 | 203.4 (51.6)
  Cycle 13, Day 1: number analyzed (Participants) | 74
  Cycle 13, Day 1 | 222.8 (30.3)

17. Secondary Outcome: Predose Plasma Concentration (Ctrough) of Avelumab
Description: The LLQ of avelumab was 0.20 mcg/mL. Data for this outcome measure was not collected for reporting group "Best Supportive Care", since avelumab was not administered in this arm.
Time Frame: Pre-dose (0 hour) on Day 1 of Cycle 1, 2, 3, 5, 7, 9, 11, 13 and Day 15 of Cycle 1, 2, 3 (each cycle=28 days)
Population: Avelumab PK parameter analysis set: all participants who received at least one dose of avelumab and who had at least one post-dose concentration measurement above the LLQ for avelumab. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'n' signifies participants evaluable for this OM at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Avelumab + Best Supportive Care (BSC)
Number analyzed (Participants) | 344
microgram per milliliter (mcg/mL)
  Cycle 1, Day 1: number analyzed (Participants) | 321
  Cycle 1, Day 1 | 3.1 (247.6)
  Cycle 1, Day 15: number analyzed (Participants) | 296
  Cycle 1, Day 15 | 22.2 (48.6)
  Cycle 2, Day 1: number analyzed (Participants) | 268
  Cycle 2, Day 1 | 25.2 (64.2)
  Cycle 2, Day 15: number analyzed (Participants) | 253
  Cycle 2, Day 15 | 26.5 (65.4)
  Cycle 3, Day 1: number analyzed (Participants) | 240
  Cycle 3, Day 1 | 26.4 (76.2)
  Cycle 3, Day 15: number analyzed (Participants) | 220
  Cycle 3, Day 15 | 25.7 (85.2)
  Cycle 5, Day 1: number analyzed (Participants) | 183
  Cycle 5, Day 1 | 26.8 (67.5)
  Cycle 7, Day 1: number analyzed (Participants) | 146
  Cycle 7, Day 1 | 29.7 (60.2)
  Cycle 9, Day 1: number analyzed (Participants) | 111
  Cycle 9, Day 1 | 32.4 (55.9)
  Cycle 11, Day 1: number analyzed (Participants) | 90
  Cycle 11, Day 1 | 29.8 (68.9)
  Cycle 13, Day 1: number analyzed (Participants) | 75
  Cycle 13, Day 1 | 32.4 (54.9)

18. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Avelumab by Never and Ever Positive Status
Description: ADA against avelumab in serum samples was determined and reported separately for ADA never positive and ADA ever positive participants. Participants were considered ADA ever-positive if they had at least one positive ADA result at any time point during study and were otherwise considered negative. Data for this outcome measure was not planned to be collected and analyzed for reporting arm "Best Supportive Care", since avelumab was not administered in this arm.
Time Frame: From randomization up to the 30-Day Follow-up visit (maximum duration of up to approximately 68 months)
Population: The immunogenicity analysis set included all participants who had received at least one dose of study drug and who had at least one ADA sample collected for avelumab in the avelumab containing arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Best Supportive Care (BSC)
Number analyzed (Participants) | 344
Participants
  Never-positive | 278
  Ever-positive | 66

19. Secondary Outcome: Number of ADA Ever Positive Participants For Each Serum of ADA Titers for Avelumab
Description: Serum samples were assayed for ADA using a validated analytical method. Number of ADA ever positive participants for each serum of ADA titer (60, 180, 540, 1620, 4860, 14580, and 131220) are reported.
Time Frame: From randomization up to the 30-Day Follow-up visit (maximum duration of up to approximately 68 months)
Population: The immunogenicity analysis set included participants who had received at least one dose of study drug and who had ADA ever-positive results. Here "Overall number of participants analyzed" signifies participants who had data available for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Best Supportive Care (BSC)
Number analyzed (Participants) | 66
Participants
  60 | 4
  180 | 14
  540 | 19
  1620 | 10
  4860 | 11
  14580 | 7
  131220 | 1

20. Secondary Outcome: Number of Participants With Neutralizing Antibodies (nAb) Against Avelumab by Never Positive and Ever Positive Status
Description: nAb against avelumab in serum samples was determined and reported separately for nAb never positive and nAb ever positive participants. Participants were considered nAb ever-positive if they had at least one positive nAb result at any time point during study and were otherwise considered negative.
Time Frame: From randomization up to the 30-Day Follow-up visit (maximum duration of up to approximately 68 months)
Population: The immunogenicity analysis set included all participants who had received at least one dose of study drug and who had at least one nAb sample collected for avelumab in the avelumab containing arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Best Supportive Care (BSC)
Number analyzed (Participants) | 344
Participants
  Never-positive | 284
  Ever-positive | 60

21. Secondary Outcome: Number of Participants With Programmed Death Receptor-1 Ligand 1 (PD-L1) Biomarker Expression in Tumor Tissue as Assessed by Immunohistochemistry (IHC)
Description: PD-L1 assessment was performed using immunohistochemistry on pre-treatment tumor tissue samples. Participants were classified as having PD-L1 -positive status if at least one of the following three criteria were met: at least 25% of tumor cells stained for PD-L1, at least 25% of immune cells stained for PD-L1 if more than 1% of the tumor area contained immune cells, or 100% of immune cells stained for PD-L1 if no more than 1% of the tumor area contained immune cells.
Time Frame: Up to 41 months at the time of the analysis
Population: The full analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
Participants
  Positive | 189 | 169
  Negative | 139 | 131
  Unknown | 22 | 50

22. Secondary Outcome: Number of Participants With Cluster of Differentiation 8 (CD8) T Lymphocytes (Cytotoxic T Lymphocytes)
Description: Number of Participants With CD8 T Lymphocytes (Cytotoxic T lymphocytes) were presented in this outcome.
Time Frame: Up to approximately 60 months
Population: Biomarker analysis set is a subset of the safety analysis set and included participants who have at least one baseline biomarker assessment performed. Here, 'Overall Number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 337 | 326
Participants | 148 | 134

23. Secondary Outcome: Change From Baseline in National Comprehensive Cancer Network- Functional Assessment of Cancer Therapy (NCCN-FACT) Bladder Symptom Index- 18 (FBlSI-18) Score at Day 1 of Cycle 6
Description: NCCN-FACT FBlSI-18 is an 18-item participant completed questionnaire, designed to assess impact of cancer therapy on urothelial cancer-related symptoms and quality of life based on numerical point scoring of symptoms/concerns. It included four subscales: Disease related symptoms- physical subscale with 9 items, disease related symptoms- emotional subscale with 2 items, treatment side effects subscale with 5 items and general function/well-being subscale with 2 items. Participants rated their level of symptoms for each item using 5-point scale ranging from 0=not at all to 4=very much. Items that were negatively framed, and the scores were reversed for analysis so that higher scores= good quality of life. Overall score: total of 18 items, ranging from 0=severely symptomatic to 72=asymptomatic. Higher scores= better functioning or lower symptom burden.
Time Frame: Baseline, Day 1 of Cycle 6 (1 cycle=28 days)
Population: The full analysis set included all randomized participants. Here, 'Overall number of participants analyzed' signifies participants who had data available for this outcome measure and 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 332 | 329
units on a scale
  Baseline | 53.3 (9.59) | 52.7 (9.31)
  Change at Day 1 of Cycle 6: number analyzed (Participants) | 178 | 109
  Change at Day 1 of Cycle 6 | 1.0 (8.25) | 1.6 (8.35)

24. Secondary Outcome: Time to Deterioration (TTD) Based on National Comprehensive Cancer Network- Functional Assessment of Cancer Therapy (NCCN-FACT) Bladder Symptom Index- 18 (FBlSI-18) Disease Related Symptoms-Physical Subscale (DRS-P) Scores
Description: NCCN-FACT FBlSI-18: an 18-item participant completed questionnaire, designed to assess impact of cancer therapy on urothelial cancer-related symptoms and quality of life based on numerical point scoring of symptoms/concerns. It included four subscales: Disease related symptoms-physical subscale with 9 items, disease related symptoms-emotional subscale with 2 items, treatment side effects subscale with 5 items, general function/well-being subscale with 2 items. Participants rated their level of symptoms for each item using 5-point scale ranging: 0=not at all to 4=very much. For items negatively framed, scores were reversed for analysis so that higher scores= good quality of life. DRS-P score: total 9 items, ranging from 0=severely symptomatic to 36= asymptomatic. Higher scores=better functioning or lower symptom burden. TTD: time from randomization to first time participant's score showed 3 point or greater decrease from baseline in FBlSI-DRS-P subscale for 2 consecutive assessments.
Time Frame: From randomization up to the 90-Day Follow-up Visit (maximum duration of up to 41 months)
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 350 | 350
months | NA [13.9 to NA] — Median and upper limit of 95% CI were not estimable due to the small number of events. | 13.8 [12.9 to NA] — The upper limit of 95% CI was not estimable due to the small number of events.
Statistical Analysis 1: Comparison: Avelumab + Best Supportive Care (BSC) vs Best Supportive Care; Test type: Superiority; p = 0.9130, Log Rank; Cox Proportional Hazard = 1.26, 95% CI 1-sided [lower limit 0.901]

25. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Overall Health Utility Score at Cycle 6
Description: The EQ-5D-5L was a 6-item participant-completed questionnaire designed to assess health status in terms of a single utility score. There were 2 components to the EQ-5D-5L, a Health State Profile which had individuals rate their level of problems (none, slight, moderate, severe, extreme/unable) in 5 areas (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), and a Visual Analogue Scale (VAS) in which participant rated their overall health status from 0 (worst imaginable) to 100 (best imaginable). Published UK weights was used to create a single summary utility score. Utility scores range from -0.594 to 1, with low scores representing lower health status.
Time Frame: Baseline, Day 1 of Cycle 6 (1 cycle=28 days)
Population: The full analysis set included all participants who were randomized. Here, 'Overall number of participants analyzed' signifies participants who had data available for this outcome measure and 'number analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 336 | 327
units on a scale
  Baseline | 0.814 (0.1794) | 0.792 (0.2013)
  Change at Day 1 of Cycle 6: number analyzed (Participants) | 181 | 111
  Change at Day 1 of Cycle 6 | -0.029 (0.1919) | -0.020 (0.1684)

26. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) - Visual Analog Scale (VAS) Score at Cycle 6
Description: The EQ-5D-5L was a 6-item participant-completed questionnaire designed to assess health status in terms of a single utility score. There were 2 components to the EQ-5D-5L, a Health State Profile which had individuals rate their level of problems (none, slight, moderate, severe, extreme/unable) in 5 areas (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), and a Visual Analogue Scale (VAS) in which participant rated their overall health status from 0 (worst imaginable) to 100 (best imaginable), higher scores indicating a better health state.
Time Frame: Baseline, Day 1 of Cycle 6 (1 cycle=28 days)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
Number analyzed (Participants) | 335 | 325
units on a scale
  Baseline | 74.9 (18.87) | 74.9 (16.34)
  Change at Day 1 of Cycle 6: number analyzed (Participants) | 183 | 109
  Change at Day 1 of Cycle 6 | 1.6 (17.74) | 0.2 (14.74)

ADVERSE EVENTS:
Time Frame: For ''Avelumab + Best Supportive Care (BSC)'' reporting group: Day 1 up to 90 days after last dose of study drug and for ''Best Supportive Care'' reporting group: Day 1 up to 90 days after end of treatment visit, for a maximum duration of up to 70 months for both groups.
Description: Same event may appear as both non-SAE and Serious Adverse Events (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. All-Cause Mortality, SAEs and non-SAEs were assessed in Safety Analysis set.
Arm/Group | Avelumab + Best Supportive Care (BSC) | Best Supportive Care
All-Cause Mortality (participants affected / at risk) | 225/344 | 242/345
Serious Adverse Events (participants affected / at risk) | 111/344 | 73/345
Other Adverse Events (participants affected / at risk) | 321/344 | 214/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Best Supportive Care (BSC) (N=344) | Best Supportive Care (N=345)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Disease progression (General disorders) | 4 | 16
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Mass (General disorders) | 0 | 1
Pain (General disorders) | 4 | 1
Pyrexia (General disorders) | 2 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cellulitis orbital (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Gallbladder abscess (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 4 | 4
Pyelonephritis acute (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 4 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 17 | 7
Urosepsis (Infections and infestations) | 1 | 2
Vascular device infection (Infections and infestations) | 2 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Stomal hernia (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Device occlusion (Product Issues) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 6
Anuria (Renal and urinary disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 5 | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 4 | 1
Immune-mediated nephritis (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Cystocele (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Best Supportive Care (BSC) (N=344) | Best Supportive Care (N=345)
Anaemia (Blood and lymphatic system disorders) | 47 | 22
Hyperthyroidism (Endocrine disorders) | 21 | 1
Hypothyroidism (Endocrine disorders) | 44 | 2
Asthenia (General disorders) | 64 | 19
Chills (General disorders) | 29 | 3
Fatigue (General disorders) | 66 | 23
Influenza like illness (General disorders) | 20 | 4
Oedema peripheral (General disorders) | 24 | 21
Pyrexia (General disorders) | 56 | 12
Abdominal pain (Gastrointestinal disorders) | 34 | 23
Constipation (Gastrointestinal disorders) | 60 | 34
Diarrhoea (Gastrointestinal disorders) | 63 | 17
Nausea (Gastrointestinal disorders) | 55 | 22
Vomiting (Gastrointestinal disorders) | 45 | 12
Influenza (Infections and infestations) | 23 | 11
Nasopharyngitis (Infections and infestations) | 33 | 13
Upper respiratory tract infection (Infections and infestations) | 24 | 8
Urinary tract infection (Infections and infestations) | 53 | 33
Infusion related reaction (Injury, poisoning and procedural complications) | 30 | 0
Alanine aminotransferase increased (Investigations) | 19 | 3
Amylase increased (Investigations) | 24 | 3
Blood creatine phosphokinase increased (Investigations) | 18 | 2
Blood creatinine increased (Investigations) | 29 | 6
Lipase increased (Investigations) | 22 | 1
Decreased appetite (Metabolism and nutrition disorders) | 48 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 68 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 57 | 34
Myalgia (Musculoskeletal and connective tissue disorders) | 32 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 23
Dizziness (Nervous system disorders) | 23 | 12
Headache (Nervous system disorders) | 27 | 9
Insomnia (Psychiatric disorders) | 24 | 9
Haematuria (Renal and urinary disorders) | 38 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 49 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 23 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 64 | 6
Rash (Skin and subcutaneous tissue disorders) | 43 | 5
Hypertension (Vascular disorders) | 22 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT02603432/Prot_002.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT02603432/SAP_001.pdf